CLINICAL TRIAL: NCT04012320
Title: Efficacy and Safety on the Use of Bisphosphonates in Paediatrics
Acronym: Bisphosphonate
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2018/TAT-01
Record Dates: First submitted 2019-06-14; First posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Bone Fragile; Bisphosphonate-Associated Osteonecrosis; Children; Adverse Events
MeSH Terms: conditions — Bisphosphonate-Associated Osteonecrosis of the Jaw | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pamidronate therapy
  Interventions: Other: No intervention, observational study
- Zoledronate therapy
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study — No intervention, observational study

SUMMARY:
The investigators suppose that the impact of bisphosphonate therapy is beneficial on the bone during the growth period with few adverse events.

ELIGIBILITY:
Inclusion Criteria:

* be under 18 years of age
* have been treated by intravenous bisphosphonates for primary or secondary osteoporosis

Exclusion Criteria:

* be over 18 years of age

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients under 18 years old who started intravenous bisphosphonates for primary or secondary osteoporosis in paediatric departments of Montpellier and Nimes University Hospitals between January 2012 and August 2018 were included.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
fracture rates | 2 years
  (numbers)
bone mineral density | 2 years
  (Z-score)
pain frequency | 2 years
  (never, occasional, regular)

CONTACTS AND LOCATIONS:
Locations (1):
- CHUNimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: Undecided